CLINICAL TRIAL: NCT04249375
Title: Integrating Pediatric Pharmacogenomic Testing Into the Canadian Health Care System
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Genome Canada (Other); Dynacare Laboratories, Inc. (Unknown)
Responsible Party: Principal Investigator, Bruce Carleton, Director, Pharmaceutical Outcomes Programme, University of British Columbia
Other Study IDs: H18-01383
Record Dates: First submitted 2019-09-24; First posted 2020-01-30 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Adverse Drug Reaction (ADR)
Keywords: Pharmacogenomics; Pediatrics; Adverse Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA samples will be retained for genomic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project addresses the problem of adverse drug reactions in the three most frequently prescribed therapeutic classes of drugs in children: antibiotics, analgesics, and mental health medications.

We will conduct pilot testing of a pharmacogenomic testing panel and study how the tests and generated test results are utilized and understood by physicians, pharmacists, patients and their families.

DETAILED DESCRIPTION:
The specific objectives are to:

1. Implement a pilot pharmacogenomics program to test medication safety and effectiveness of antibiotics, analgesics and mental health medication to enhance prescribing decision-making.
2. Develop data collection forms to collect necessary patient information from the prescribing physicians.
3. Develop pharmacogenomics reports to return results to physicians, pharmacists, patients and their families.
4. Determine how the tests and results are perceived and utilized by physicians, pharmacists, patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be enrolled if they can benefit from pharmacogenomic testing. This means their physician is considering the use of a drug that is part of the panels (analgesics, antibiotics, and mental health medication) or they are already using one.

Exclusion Criteria:

* Patients who do not speak or understand English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any individual who is currently on an analgesic, antibiotic and/or mental health medication that is part of the panels.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
150 participants on analgesics, anti-infectives and psychotropics will be given pharmacogenomic recommendations for the risk of gene related adverse events prior to or during treatment. | June 2020
  We will be able to determine the barriers and facilitators of the implementation of the pharmacogenomic service in a health care facility.
  This will be done by using standardized questionnaires after each pharmacogenomic report is issued. The prescriber and the patient will both answer questions about the utility of the genetic results, the format of the report and the clarity of the content.
  Results will be recorded and summarized every 25 patients in order to improve the service and the recommendations through the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.cpnds.ubc.ca